CLINICAL TRIAL: NCT07160946
Title: Research on Risk Assessment and Intervention of HBV-Related Liver Cancer Based on Multimodal Data Fusion
Brief Title: Risk Assessment for HBV-Related Liver Cancer
Status: Recruiting | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Lin Bingliang, Prof., Sun Yat-sen University
Other Study IDs: Spark Liver Health
Record Dates: First submitted 2025-08-02; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-07

CONDITIONS: HBV-related Liver Cirrhosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Routine follow-up group: Patients in this cohor will be followed up every 24 weeks (or every 8-12 weeks for extremely high-risk population) routinely. Alpha fetoprotein, PIVKA-II, liver imaging examination, liver function, et al will be performed for these patients at each follow-up point.
- AI system follow-up group: Patients in this cohor will be followed up every 24 weeks (or every 8-12 weeks for extremely high-risk population). Alpha fetoprotein, PIVKA-II, liver imaging examination, liver function, et al will be performed for these patients at each follow up point. An AI system will be used to manage follow-up patients.
  Interventions: Other: AI folow-up system

INTERVENTIONS:
Other: AI folow-up system — In AI follow-up group, patients will be followed up by an AI system.
  Groups: AI system follow-up group

SUMMARY:
Liver cancer is a severe disease worldwide. The incidence and mortality rates of liver cancer in China is the highest in the world. This project aims to perform a prospective, multi-center, large sample cohort study for HBV related high-risk individuals. Based on multimodal data fusion and AI technique, stratified management and follow-up system are conducted for HBV-related high-risk populations of liver cancer, in order to improve the early diagnosis rate of liver cancer.

ELIGIBILITY:
Inclusion Criteria: must meet (a) and any one of (b) to (g).

* (a).Positive for Hepatitis B surface antigen; (b).Ultrasound/CT/MR indicates liver cirrhosis; (c). Type II diabetes; (d). Has family history of liver cirrhosis/ liver cancer; (e). Long term alcohol consumption history (>5 years), equivalent to alcohol consumption of ≥ 40g/d for males and ≥ 20g/d for females; (f). Liver histology Metavir fibrosis score F3 or above; (g). Fibroscan value (LSM) ≥ 8.0kPa.

Exclusion Criteria:

* (a).Diagnosed with malignant tumors; (b). Post liver transplantation; (c). Infected with HIV; (d). Expected survival time<1 year; (e). With marked organ dysfunctions(heart, brain, kidney, lung, endocrine system, blood, etc.) or psychiatric patients.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The diagnostic rate of stage I liver cancer in China (AJCC-7 TNM staging system) is 17.5%. It is planned to increase the diagnostic rate of stage I liver cancer by 50% through this project, reaching 26.3%, power=0.9, a=0.05. PASS software calculated that a total of 958 liver cancer patients need to be enrolled in both groups. It is known that the annual incidence of liver cancer in patients with hepatitis B cirrhosis is 3% -6%. If calculated by 4%, it is estimated that the patients will be enrolled in one year, followed up for five years, and the lost rate is 10%, 5470 patients will need to be enrolled. Ultimately, this study plans to enroll 6000 patients.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2025-05-10 (Actual); Primary Completion 2032-12-30 (Estimated); Study Completion 2032-12-30 (Estimated)

PRIMARY OUTCOMES:
Number and specific time of participants progressing to liver cancer | 5 years
  Number and specific time of participants progressing to liver cancer

SECONDARY OUTCOMES:
Survival time | 5 years
  Participants' survival time after being diagnosed with liver cancer.

OTHER OUTCOMES:
Incidence of adverse events for the participants | 5 years
  Incidence of ascite, hepatorenal system, hepatic encephalopathy, gastrointestinal bleeding, etc. for all the participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Third Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Shan T, Ran X, Li H, Feng G, Zhang S, Zhang X, Zhang L, Lu L, An L, Fu R, Sun K, Wang S, Chen R, Li L, Chen W, Wei W, Zeng H, He J. Disparities in stage at diagnosis for liver cancer in China. J Natl Cancer Cent. 2023 Jan 3;3(1):7-13. doi: 10.1016/j.jncc.2022.12.002. eCollection 2023 Mar. PMID 39036312
- [Background] Singh SP, Madke T, Chand P. Global Epidemiology of Hepatocellular Carcinoma. J Clin Exp Hepatol. 2025 Mar-Apr;15(2):102446. doi: 10.1016/j.jceh.2024.102446. Epub 2024 Oct 28. PMID 39659901
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/39659901/